CLINICAL TRIAL: NCT01622842
Title: Bioimpedance of Human Tissue of the Upper Arm and Arterial Distension
Brief Title: Bioimpedance and Arterial Distension
Acronym: SenseC1
Status: Completed | Type: Observational
Sponsor: Sense A/S (Industry)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: H-1-2011-076
Record Dates: First submitted 2012-06-08; First posted 2012-06-19 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: Impedance; Electrical; Tissue; Excitation frequency; arterial distension; distension wave form
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bioimpedance: 8 females and 8 males BMI from 19 to 46 SBP from 119 to 182

SUMMARY:
The overall objectives were to investigate if characteristic dimensions for tissue and vessels determined from measured bioimpedance spectra would provide the same values as dimensions determined from MR images of the upper arm and verify that temporal variations of impedances could be converted to blood pressure.

DETAILED DESCRIPTION:
It is emphasized that measurements of pulse wave velocity was not a part of this trial, which implies that only uncalibrated blood pressures could be measured. The specific objectives were:

1. To determine conductivities and permittivities in the spectral region from 1 KHz to 1 MHz for persons with: (a) a normal distribution of fat and muscles, (b) exceptionally thick layers of subcutaneous fat, and (c) exceptionally thin layers of subcutaneous fat. Both sexes should be represented.
2. To verify that temporal variations synchronous with the heartbeat could be measured on all three groups.

Hypotheses:

A. That experimentally in vivo determined electrical parameters for tissues would differ considerably from theoretical values and from values measured in vitro experiments.

B. That the variations of the electrical parameters would exhibit little variation from person to person.

C. Those simple experimental relations can be established for the electrical parameters by including a simple vascularization model.

D. That it is possible to measure temporal variation of the impedance, which are synchronous with the heartbeat.

E. That the measured values would facilitate the calculation of the differential blood pressure with accuracies better than 10 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years
* Mental ability to understand information to test subjects

Exclusion Criteria:

* Serious illness
* Allergic reactions to ECG or EMG electrodes
* Mentally unstable or unable to perceive instructions
* Metal implants
* Claustrophobia
* Disqualified for MR scanning
* Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Equal number of females and males. Large variations of BMI Large variations of BP
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Conductivities and permittivities in the spectral region from 1 KHz to 1 MHz. | 1 hour
  Measured on persons with: (a) a normal distribution of fat and muscles, (b) exceptionally thick layers of subcutaneous fat, and (c) exceptionally thin layers of subcutaneous fat. Both sexes should be represented. Muscles and vessels followed expectations based on litterature values for electrical properties. Subcutaneous fat had a higher conductivity and permittivity than predicted from literature values in all cases.

SECONDARY OUTCOMES:
Temporal variations synchronous with the heartbeat | 1 hour
  The temporal variations of impedances measured on persons with: (a) a normal distribution of fat and muscles, (b) exceptionally thick layers of subcutaneous fat, and (c) exceptionally thin layers of subcutaneous fat. Both sexes should be represented. Temporal variations could be measured on all three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lading, Prof., Study Director — Sense A/S; Tine W Hansen, MD, PhD, Principal Investigator — Rigshospitalet (Copenhagen Univ. Hospital)
Locations (1):
- Rigshopsitalet (Copenhagen Univ. Hospital), Copenhagen, Denmark